CLINICAL TRIAL: NCT05573685
Title: A Randomized, Controlled, Single-Blind, Exploratory Basket Study to Evaluate the Effects of a DiNaMo™ Component Training in Adults With Chronic Pain-Related Disorders
Brief Title: Basket Study (CT-100-002) to Evaluate the Effects of a DiNaMo™ Component Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CT-100-D-002
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis; Diabetic Neuropathy; Fibromyalgia; Irritable Bowel Syndrome
Keywords: Smartphone, RA, diabetic neuropathy, fibromyalgia, IBS
MeSH Terms: conditions — Arthritis, Rheumatoid; Diabetic Neuropathies; Fibromyalgia; Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single blind, randomized into 3:1 ratio (3 DiNaMo Study Apps of 4 indications: 1 Digital Control App)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DiNaMo Study App (Active Comparator): Randomization ratio as 3 DiNaMo Study Apps: 1 Digital Control App
  Interventions: Device: DiNaMo Study App
- Digital Control App (Placebo Comparator): Randomization ratio as 3 DiNaMo Study Apps: 1 Digital Control App
  Interventions: Device: Placebo App

INTERVENTIONS:
Device: DiNaMo Study App — Study App to be used in patients with 1 of the 4 indications of rheumatoid arthritis, fibromyalgia Irritable Bowel Syndrome, Diabetic Neuropathy
  Arms: DiNaMo Study App
Device: Placebo App — Placebo App to be used in patients with 1 of the 4 indications of rheumatoid arthritis, fibromyalgia Irritable Bowel Syndrome, Diabetic Neuropathy
  Arms: Digital Control App

SUMMARY:
CT-100 is a platform that provides interactive, software based therapeutic components that may be used as part of a multimodal treatment in supplementary or standalone prescription or nonprescription software-based digital therapeutics (PDT/DTx), being developed by Click Therapeutics, Inc. (Click).

DETAILED DESCRIPTION:
The Study App (CT-100-002) contains a class of Digital Neuro-activation and Modulation (DiNaMo™) mechanisms of action that are part of the Click Neurobehavioral Intervention (CNI) Platform™. DiNaMo™ provide interactive, software based therapeutic components that may be included in a multimodal treatment for developing future digital therapeutics.

Chronic pain is a transdiagnostic condition which manifests in patients with diverse underlying pathologies such as rheumatoid arthritis, diabetic neuropathy, fibromyalgia, and irritable bowel syndrome. This basket study aims to evaluate the efficacy, safety, and tolerability of CT-100-002 on measures of pain, pain-related functioning, and mood across multiple indications. The study results will further future clinical development of digital therapeutics comprising DiNaMo™ mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Meets indication-specific eligibility criteria as reported by the study participant with adequate clinical documentation
* Self-reported average pain intensity during the last 7 days of ≥ 3 of 10 on the Numeric rating Scale (NRS scale) associated with the primary indication
* Fluent in written and spoken English (confirmed by ability to read and comprehend the informed consent form.)
* Willing and able to comply with study protocol and assessments, evidenced by completion of the Screening Survey.
* Lives in the United States.
* Has an active email address and is willing and able to receive email messages.
* Is the sole user of an iPhone with iPhone operating systems (iOS) 14 or later capabilities or a smartphone with an Android operating system (OS) 10 or later capabilities with cellular and/or internet access for the duration of the study period.

Exclusion Criteria:

* Has a comorbid acute pain condition, such as from current injuries
* Participation in a clinical trial (including psychotherapy, mindfulness, cognitive training, or drug treatment) within the last 2 months
* Initiation or change in primary disease-specific medication for 30 days prior to entering the study
* Self-reported substance use disorder within the past 1 year
* Daily use of opioids of 30 MME (Morphine Milligram Equivalents) or more
* Substance use disorder within the past 1 year.
* Initiation or change in central nervous system-active medication (e.g., antidepressants) during the last 2 months.
* Participation in a clinical trial within the last 2 months.
* Planning to introduce new therapies or change therapies during the study duration
* Visual, dexterity or cognitive deficit so severe that precludes the use of an app per investigator judgment.
* Severe psychiatric disorder involving a history of psychosis
* Other significant medical condition that may confound the interpretation of findings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
To estimate the effect size for changes in pain experience (interference) in the Treatment App group compared to the Digital Control App group | Change from Baseline to Week 4
  Effect size change as measured by the Numerical Rating Scale (NRS) questionnaire, from the lowest (0) to the highest (10)

SECONDARY OUTCOMES:
To explore the feasibility of remote digital DiNaMo training Study App in participants with chronic pain | User experience questionnaire of feasibility recorded on baseline and Week 4
  Feasibility is measured by using User Experience Questionnaire including engagement and experience with the Study App in participants with chronic pain as measured by metrics such as daily app usage and daily time in the app. The questionnaire will ask questions related to the perceived enjoyment, challenges, and related user experience.
To estimate the effect size for changes in attention to pain in the Treatment App group compared to the Digital Control App group | Change from baseline to Week 4
  Change is measured by the Pain Vigilance and Awareness Questionnaire (PVAQ), from the lowest (0) to the highest (5).
To estimate the effect size for changes in pain catastrophizing in the Treatment App group compared to the Digital Control App group | Change from baseline to Week 4
  Change is measured by the Pain Catastrophizing Scale (PCS) from the lowest (0) to the highest (4).
To estimate the effect size for changes in confidence in dealing with chronic pain in the Treatment App group compared to the Digital Control App group | Change from baseline to Week 4
  Change is measured by the Pain Self-efficacy Questionnaire (PSEQ) from the lowest (0) to the highest (6).

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MD, PhD, FAAN, Principal Investigator — Click Therapeutics, Inc.
Locations (1):
- Click Therapeutics, New York, New York, United States